CLINICAL TRIAL: NCT03038009
Title: Evaluation of the Efficacy and Safety of Different Duration of Proton Pump Inhibitor for Prevention of Upper Gastrointestinal Mucosal Injury in Patients Taking 12-month Dual Antiplatelet Therapy After Coronary Artery Bypass Graft Surgery
Brief Title: Proton Pump Inhibitor Prevent Dual Antiplatelet Agents Induced Gastrointestinal Ulcer After Coronary Artery Bypass Graft
Acronym: DACAB-GI-2
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: A new registration has been submitted due to a redesign of the study protocol.
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Lifen YU, Associate Professor, Department of Gastroenterology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IISR-2016-101603
Record Dates: First submitted 2017-01-29; First posted 2017-01-31 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Gastric Ulcer Induced by Antiplatelet Agent; Ulcer of the Gastrointestinal Tract; Proton Pump Inhibitor
Keywords: Coronary Artery Bypass Graft; Dual Antiplatelet Therapy; Gastrointestinal; Mucosal Injury; Proton Pump Inhibitor
MeSH Terms: conditions — Peptic Ulcer | interventions — Pantoprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-month therapy (Active Comparator): Pantoprazole, 40mg, tablet, oral, once daily for 1 month.
  Interventions: Drug: Pantoprazole
- Twelve-month therapy (Experimental): Pantoprazole, 40mg, tablet, oral, once daily for 12 months.
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — Pantoprazole (40mg qd) will be concomitant used with DAPT
  Other Names: PANTOLOC, Tablet from Takeda Pharmaceutical Company Limited

SUMMARY:
The purpose of this study is to determine whether 12-month prophylactic treatment with pantoprazole is superior to 1-month therapy without major cardiovascular events (MACE) increased significantly, in prevention of dual antiplatelet therapy (DAPT)-induced upper gastrointestinal (GI) mucosal injury after coronary artery bypass graft (CABG) surgery. The potentially serious harm of DAPT on gastroduodenal mucosa will be assessed by esophagogastroduodenoscopy (EGD).

DETAILED DESCRIPTION:
Endoscopic evaluation of gastroduodenal mucosal injury:

Based on the modified Lanza score, the new endoscopic evaluation system established in the DACAB-GI-1 study includes 6 grades of mucosal injuries. Grade 0: normal mucosa; Grade 1: erythema or petechiae only; Grade 2: 1 to 2 erosive lesions; Grade 3: 3 to 10 erosive lesions; Grade 4: more than 10 erosive lesions or small ulcers (diameter: 3-5mm); Grade 5: an ulcer is greater than 5 mm in diameter. Comprehensive results of gastroduodenal mucosal injury will be marked as G0-5 (G: gastro) and D0-5 (D: duodeno) together. Mild injury was defined as level II or less. Severe injury was defined from level III to V, which should be treated with proton pump inhibitor (PPI) to decrease the risk of upper GI bleeding. The new level system is as following: Level 0: G0D0; Level I: G1D0-1/G0D1; Level II: G2D0-2/G0-1D2; Level III: G3D0-3/G0-2D3; Level IV: G4D0-4/G0-3D4; Level V: G5D0-5/G0-4D5.

Sample size justification:

Until now, no published data or reference is available for the efficacy of pantoprazole when concomitant use with DAPT. The results from the preliminary study (DACAB-GI-1) showed that the percentage of serious gastroduodenal mucosal lesions (Level III-V) in patients treated with PPIs for 1, 3 and more than 6 months were 36.76%, 28.45% and 17.65%, respectively. Therefore, the efficacy difference of pantoprazole is estimated to be 18% between 2 groups. The average incidence of gastroduodenal mucosal injury is estimated to be 36% in the control group (1-month therapy of pantoprazole), and the corresponding incidence in the experimental group (12-month therapy of pantoprazole) is estimated to be 18%.

The determination of minimal sample size is as following: Group sample sizes of 93 in the experimental group and 93 in the control group achieve 80% power to detect a difference between the group proportions of -18%. The proportion in the experimental group is assumed to be 36% under the null hypothesis and 18% under the alternative hypothesis. The proportion in the control group is 36%. The test statistic used is Pearson Chi-Squared test. The significance level of the test was targeted at 0.05. The significance level actually achieved by this design is 0.0522. Considering 10% of the lost and/or drop-out rate, the final sample size estimated will be 104 in the experimental group and control group, respectively. The total sample size is no less than 208.

ELIGIBILITY:
Inclusion Criteria:

Each patient should meet all of the inclusion criteria and none of the exclusion criteria for this study:

1. Provision of informed consent prior to any study specific procedures.
2. CABG surgery is performed for the first time.
3. Need 12-month DAPT (aspirin 100mg qd plus clopidogrel 75mg qd or aspirin 100mg qd plus ticagrelor 90mg bid depending on randomisation) immediately following CABG surgery according to the guideline.
4. Concomitant use of pantoprazole (40mg qd) for at least 1 moth following CABG surgery.
5. Willing to undergo EGD twice a year (at 6th and 12th month following CABG surgery, respectively).
6. Willing to undergo 13C-UBT prior to CABG surgery.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled.

1. History of previous active peptic ulcer within 3 months prior to enrollment.
2. Planned use of PPI to treat gastric-acid associated diseases (e.g. gastroesophageal reflux disease, GERD)
3. Contraindications for aspirin, clopidogrel, ticagrelor and pantoprazole use (e.g. known allergy)
4. Anticipated concomitant oral or intravenous therapy with strong cytochrome P450 3A4 (CYP3A4) inhibitors or CYP3A4 substrates with narrow therapeutic indices, that cannot be stopped for the course of the study.

   * Strong inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir
   * CYP3A4 substrates with narrow therapeutic index: quinidine, simvastatin at doses > 40mg daily or lovastatin at doses > 40mg daily.
5. Need for chronic oral anticoagulant therapy or chronic low-molecular-weight heparin.
6. History of previous intracerebral bleeding at any time, GI bleeding within the past 3 months prior to enrollment, or major surgery within 30 days prior to enrollment.
7. Known moderate to severe liver disease (e.g. gastroesophageal varices, ascites and/ or clinical signs of coagulopathy)
8. Renal failure requiring dialysis.
9. Women of child-bearing potential who are not willing to use a medically accepted method of contraception that is considered reliable in the judgement of investigator OR women who have a positive pregnancy test at enrolment or randomisation OR women who are breasting-feeding.
10. Inability of patient to understand and/or comply with study procedures and/or follow up, in the opinion of the investigator, OR any conditions that, in the opinion of the investigator, many render the patient unable to complete the study.
11. Any condition which in the opinion of the investigator would make it unsafe or unsuitable for the patient to participate in this study (eg, long-term concomitant treatment with non-steroidal anti-inflammatory drugs [NSAIDs]), or any condition outside the atherothrombotic study area with a life expectancy of less than 2 years based on investigator's judgement.
12. Paticipation in another clinical study with an investigational product within 28 days prior to enrolment or previous randomization to an investigational product in another ongoing clinical study. Participation in any previous study with clopidogrel or tigagrelor.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of gastroduodenal erosions and ulcers. | up to 12 months

SECONDARY OUTCOMES:
Incidence of gastroduodenal erosions and ulcers. | up to 6 months
Incidence of upper GI major bleeding according to TIMI criteria. | up to 12 months
Incidence of upper GI minor bleeding according to TIMI criteria | up to 12 months
Incidence of major cardiovascular events (MACE, composite of cardiovascular death, myocardial infarctions, or stroke). | up to 12 months
  Safety Issue: Yes
Incidence of grafts failure. | up to 12 months
  Safety Issue: Yes

CONTACTS AND LOCATIONS:
Overall Officials: Lifen Yu, MD, Ph.D, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No